CLINICAL TRIAL: NCT05103852
Title: Feasibility, Safety and Diagnostic Input of Interventional Cardiac MRI on a Series of 35 Patients With an Indication of Right Cardiac Catheterization.
Acronym: IRM Cardiaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A03145-48
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Cardiac MRI; Right Cardiac Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with right cardiac catheterization (Experimental)
  Interventions: Procedure: Cardiac MRI

INTERVENTIONS:
Procedure: Cardiac MRI — vigilant patient installed in the MRI with compatible ECG electrodes for synchronization and monitoring, blood pressure cuff for monitoring, cardiac antenna. Sterile drape over the femoral region, femoral local anesthesia, femoral venipuncture, Swan Ganz probe venous navigation (CE marking, MRI compatible at 1.5T) with balloon inflated with 2 cc of gadolinium, navigation under real time SSFP cine sequence.

SUMMARY:
The aim of this study is to evaluate the feasibility of collecting hemodynamic data from right catheterization, all anatomical, functional, flow and substrate determination data under MRI navigation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Having an indication for a diagnostic of right cardiac catheterization at the J Cartier Hospital for one of the following pathologies: dilated, restrictive cardiomyopathy, pulmonary arterial hypertension, chronic constrictive pericarditis, chronic post-embolic pulmonary heart.
* Subject affiliated or beneficiary of a social security scheme
* Patient having freely signed the informed consent.

Exclusion Criteria:

* Pregnancy (declarative, known pregnancy, any unexplained period delay in a woman of childbearing age)
* Presence of a contraindication to MRI: intraocular metallic splinter, surgical clip for cerebral aneurysm, claustrophobia, defibrillator, implanted electronic equipment) or to gadolinium chelates (anaphylactic reactions to gadolinium chelates, creatinine clearance <= 30 ml / min).
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision; Pregnant, breastfeeding or parturient woman; Hospitalized without consent.
* Patient participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in whom it is possible to collect all the hemodynamic data for right catheterization under MRI navigation | 24 hours
  Proportion of patients in whom it is possible to collect all the hemodynamic data for right catheterization under MRI navigation, as well as all the anatomical, functional, flow and substrate determination data by magnetic resonance (N / 35,%).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Jacques Cartier, Massy, France